CLINICAL TRIAL: NCT07156799
Title: Influence of Kaempferol Gel on Alkaline Phosphatase Activity and Bone Density Around Dental Implants: A Randomized Controlled Clinical Trial
Brief Title: Kaempferol Gel , Alkaline Phosphatase Activity , Bone Density Around Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Nora Abdelgawad Mohamed, Associate Professor of Oral Medicine, Periodontology and Diagnosis, Faculty of Dental Medicine for girls, Al -Azhar University, Cairo, Egypt, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMPDR-103-2F
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Peri-implant Bone Healing and Osseointegration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): kaempferol gel application and implant placement
  Interventions: Drug: Kaempferol Gel
- control group (No Intervention): implant placement with out application of kaempferol

INTERVENTIONS:
Drug: Kaempferol Gel — Local topical application of Kaempferol gel into the implant site during one-stage delayed implant placement to enhance peri-implant bone healing and osseointegration.
  Other Names: Flavinoids
  Arms: test group

SUMMARY:
Kaempferol gel was tested as a local adjunct during implant placement in 30 patients. Compared to controls, the Kaempferol group showed significantly higher ALP activity at 2 and 4 weeks and greater bone density gain after 6 months (40.73% vs. 33.21%). These findings suggest Kaempferol enhances early bone remodeling, improves peri-implant bone quality, and may allow earlier implant loading.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigated the effect of Kaempferol gel, a natural antioxidant and bone-healing compound, on dental implant healing in the maxillary posterior region. Thirty patients were divided into two groups: one received Kaempferol gel during implant placement, while the other did not.

The study measured alkaline phosphatase (ALP) activity in peri-implant crevicular fluid at 1, 2, and 4 weeks, and bone density using CBCT at baseline and 6 months. Results showed that Kaempferol significantly boosted ALP activity at 2 and 4 weeks, suggesting faster bone remodeling. At 6 months, bone density improved in both groups, but the Kaempferol group showed a greater increase (40.73% vs. 33.21%).

In conclusion, Kaempferol gel enhanced early bone healing and improved bone density around implants, indicating its potential as a cost-effective, biocompatible adjunct to accelerate osseointegration and possibly allow earlier implant loading, particularly in patients with poor bone quality.

ELIGIBILITY:
Inclusion Criteria:

* At least one missing maxillary posterior tooth with a healed ridge

Exclusion Criteria:

* Previous bone grafting at the implant site.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — more than 18 years
Enrollment: 30 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
alkaline phosphatase level | at baseline, 1,2, 4 weeks
  Change in alkaline phosphatase (ALP) activity measured in peri-implant crevicular fluid (PICF) using ELISA to evaluate early bone remodeling activity.

SECONDARY OUTCOMES:
Bone density around implants | Baseline and 6 months postoperatively
  Change in peri-implant bone density assessed by cone beam computed tomography (CBCT) at the implant site

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nora Abdelgawad, Principal Investigator — Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt
Locations (1):
- Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Cairo Governorate, Egypt